CLINICAL TRIAL: NCT02084186
Title: The Mechanism of Moxibustion in Treating Ulcerative Colitis Based on Metabonomics
Brief Title: Moxibustion for Mild and Moderate Ulcerative Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Institute of Acupuncture, Moxibustion and Meridian (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 81303033
Record Dates: First submitted 2014-03-09; First posted 2014-03-11 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2015-12

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- moxibustion group (Experimental): herb-partitioned moxibustion on bilateral Tianshu (ST25) and Shangjuxu (ST37)
  Interventions: Other: herb-partitioned moxibustion
- bran-partitioned moxibustion (Placebo Comparator): bran-partitioned moxibustion on bilateral Tianshu (ST25) and Shangjuxu (ST37)
  Interventions: Other: bran-partitioned moxibustion

INTERVENTIONS:
Other: herb-partitioned moxibustion — Ignited moxa cones are placed upon herbal cake. Herbs are smashed into powder. Every 2.8g medicine powder mix with 3g millet wine and then be pressed into herbal cakes which are 28mm in diameter and 7mm in high with a specific mould. Then the herbal cake with a moxa cone will be fixed on Tianshu and Shangjuxu.
  Arms: moxibustion group
Other: bran-partitioned moxibustion — Ignited moxa cones are placed upon bran cake. Every 2.8g bran powder mix with 3g millet wine and then be pressed into bran cakes which are 28mm in diameter and 7mm in high with a specific mould. Then the bran cake with a moxa cone will be fixed on Tianshu and Shangjuxu.
  Arms: bran-partitioned moxibustion

SUMMARY:
The purpose of this study is to determine whether moxibustion is effective to mild and moderate ulcerative colitis and the effect of moxibustion on metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnosis of UC
* Mayo ≤10
* Patients should have never received any pharmacological therapy or if they are receiving aminosalicylates and/or prednisolone (the dosage has been taken at least 4 weeks, and should be kept the same as before throughout the trial)
* Patients should have never received antibiotic, biologicals, probiotics, acetaminophen, acetamide and contraceptive.
* A written informed consent

Exclusion Criteria:

* Patients with cardiac, encephalic, hepatic, nephric, hematopoietic system, psychotic or any other serious diseases
* Pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
disease activity index (DAI) | 3 months
  Using Mayo subscore

SECONDARY OUTCOMES:
Inflammatory Bowel Disease Questionnaire (IBDQ) | 3 months
symptom score | 3 months
histomorphology observation of intestinal mucosa | 3 months
  Using the Geboes histology score
metabolic profile of intestinal mucosa, urine, plasma and serum | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Huangan Wu, Doctor, Study Director — Shanghai Institute of Acupuncture-Moxibustion and Meridian, Shanghai University of Traditional Chinese Medicine
Locations (1):
- Shanghai Institute of Acupuncture-Moxibustion and Meridian, Shanghai, China